CLINICAL TRIAL: NCT02546648
Title: PeriOperative ISchemic Evaluation-3 Trial: A Pilot Study (POISE-3)
Brief Title: PeriOperative ISchemic Evaluation-3 Trial: A Pilot Study
Acronym: POISE-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Population Health Research Institute (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: POISE3034
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2017-08

CONDITIONS: Atherosclerotic Disease; Perioperative Bleeding
MeSH Terms: interventions — Tranexamic Acid; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid vs. matching placebo (Experimental): Tranexamic Acid 1g bolus with anesthesia induction followed by 1g bolus at the start of surgical closure.
  Interventions: Drug: Tranexamic Acid; Drug: Tranexamic Acid Placebo
- Rosuvastatin vs. matching placebo (Experimental): Rosuvastatin 20 mg orally or matching placebo once per day until 30 days after surgery
  Interventions: Drug: Rosuvastatin or matching placebo

INTERVENTIONS:
Drug: Tranexamic Acid
  Other Names: Cyklokapron
  Arms: Tranexamic Acid vs. matching placebo
Drug: Tranexamic Acid Placebo
  Arms: Tranexamic Acid vs. matching placebo
Drug: Rosuvastatin or matching placebo — Subjects who are not on a statin will also be randomized to Rosuvastatin or Rosuvastatin placebo. 40mg preoperatively, followed by 20mg postoperatively (4-6 hours after surgical close) and 20mg/day for 30 days postoperatively.
  Other Names: Crestor
  Arms: Rosuvastatin vs. matching placebo

SUMMARY:
A placebo-controlled, factorial trial to assess the impact of rosuvastatin and tranexamic acid (TXA) in patients undergoing noncardiac surgery who are at risk of a perioperative cardiovascular event.

DETAILED DESCRIPTION:
The POISE-3 pilot is a randomized controlled trial of 100 patients with, or at risk of, atherosclerotic disease who are undergoing noncardiac surgery. Utilizing a partial factorial design, the POISE-3 pilot will determine the effect of rosuvastatin versus placebo and TXA versus placebo in the perioperative setting.

ELIGIBILITY:
Inclusion Criteria:

1. undergoing noncardiac surgery
2. >45 years of age
3. expected to require at least an overnight hospital admission after surgery; AND
4. have a preoperative NT-pro-BNP measurement >100 ng/mL; OR
5. if a preoperative NT-pro-BNP measurement is not available, then the patient must fulfill 1 or more of the following 5 criteria:

   * history of coronary artery disease
   * history of peripheral vascular disease
   * history of stroke
   * undergoing major vascular surgery
   * have any 3 of the following 9 risk criteria:

     * undergoing major surgery
     * history of congestive heart failure
     * history of a transient ischemic attack
     * diabetic and currently taking an oral hypoglycemic agent or insulin
     * age >70 years
     * hypertension
     * serum creatinine > 175 umol/L (>2.0 mg/dl)
     * history of smoking within 2 years of surgery
     * undergoing emergent/urgent surgery

Exclusion Criteria:

1. planned use of systemic Tranexamic Acid during surgery
2. hypersensitivity or known allergy to TXA
3. creatinine clearance <30 mL/min (MDRD)
4. history of seizure disorder
5. history of venous thromboembolism
6. acute arterial thrombosis
7. no preoperative measurement of hemoglobin
8. subarachnoid hemorrhage within the past 30 days
9. hematuria caused by diseases of the renal parenchyma
10. previously enrolled in POISE-3 pilot trial
11. not consenting to participate in POISE-3 pilot trial prior to surgery

Patients meeting any of the following criteria will be excluded from the Rosuvastatin/Placebo arm:

1. preoperative treatment with a statin or a non statin lipid lowering drug or ciclosporin during the 48 hours before surgery
2. hypersensitivity or known allergy to Rosuvastatin
3. pre-disposed factors for myopathy or rhabdomyolysis

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Postoperative intervention discontinuation | Postoperative day 1 to 30.
  Interruption of the intervention longer than 24 hours within the first 10 days postoperatively, and longer than 48 hours from postoperative day 10 to 30.
Change in hemoglobin | Postoperative day 1.
  Change in preoperative hemoglobin to the morning hemoglobin recorded on day 1 after surgery.

SECONDARY OUTCOMES:
All-cause mortality | Postoperative day 30.
Non-fatal myocardial infarction | Postoperative day 30.
A composite of vascular mortality and non-fatal: myocardial infarction, stroke, cardiac arrest, pulmonary embolus, deep venous thrombosis, life threatening bleeding, major bleeding. | Postoperative day 30.
  Event composite

OTHER OUTCOMES:
Safety Outcomes for Rosuvastatin assessed by Statin induced myopathy | Postoperative day 30.
Safety Outcomes for Tranexamic Acid assessed by Seizure, pulmonary emboli, deep venous thrombosis, vascular mortality | Postoperative day 30.
  myocardial infarction, stroke, non-fatal cardiac arrest, and cardiac revascularization procedure.

CONTACTS AND LOCATIONS:
Overall Officials: James Khan, MD, Study Chair — Hamilton Health Sciences Corporation
Locations (2):
- Canada (2):
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marcucci M, Duceppe E, Le Manach Y, Kearon C, Eikelboom JW, Pohl K, Vincent J, Darvish-Kazem S, Srinathan SK, Neary JDD, Parlow JL, Kurz A, Gross PL, Mrkobrada M, Balasubramanian K, Sessler DI, Devereaux PJ. Tranexamic acid and rosuvastatin in patients at risk of cardiovascular events after noncardiac surgery: a pilot of the POISE-3 randomized controlled trial. Pilot Feasibility Stud. 2020 Jul 21;6:104. doi: 10.1186/s40814-020-00643-9. eCollection 2020. PMID 32699643